CLINICAL TRIAL: NCT05656157
Title: Evaluation of a Clinical Decision Support System for the Treatment of Invasive Fungal Infections
Brief Title: Evaluation of a Clinical Decision Support System for Fungal Infections
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2022_001
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Invasive Fungal Infections
Keywords: invasive fungal infections; antifungal treatment; clinical decision support system
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antifungal treatment prescribed by the clinician for an invasive fungal disease
- Antifungal treatment recommended by the clinical decision support system
  Interventions: Device: Medical device

INTERVENTIONS:
Device: Medical device — Clinical decision support system
  Groups: Antifungal treatment recommended by the clinical decision support system

SUMMARY:
Invasive fungal infections are serious and frequent diseases in our hospitals, especially in intensive care units. In accordance with the institutional recommendations, it is necessary to have a clinical decision support system to support the clinicians in a rapid and optimal prescription of antifungals for invasive fungal diseases. This clinical decision support system will benefit patients but also clinicians who will gain in medical efficiency. It will also have an ethical dimension since it will guarantee optimal antifungal treatments for all patients. The purpose of the research is to define the percentage of concordance between the medical prescription and the recommendation of the clinical decision support system.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving antifungal therapy for the treatment of invasive fungal disease

Exclusion Criteria:

* Patients not receiving antifungal therapy for the treatment of invasive fungal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving antifungal therapy for the treatment of invasive fungal disease
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of concordance between the medical prescription and the recommendation of the clinical decision support system | January to september 2023

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Bienvenu, PharmD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bienvenu AL, Pradat P, Guerin C, Aubrun F, Fellahi JL, Friggeri A, Guichon C, Hernu R, Menotti J, Monard C, Paulus S, Rimmele T, Piriou V, Chidiac C, Argaud L, Leboucher G. Evaluation of first-line therapies for the treatment of candidemia in ICU patients: A propensity score analysis. Int J Infect Dis. 2020 Apr;93:15-21. doi: 10.1016/j.ijid.2020.01.037. Epub 2020 Jan 23. PMID 31982622
- [Result] Bienvenu AL, Pavese P, Leboucher G, Berger P, Roux S, Charmillon A, Foroni L, Menotti J, Lebeaux D, Mayan R, Mondain V, Robin C, Lesprit P, Alfandari S, Kerneis S. Practical checklist for implementation of antifungal stewardship programmes. J Med Microbiol. 2022 Jun;71(6). doi: 10.1099/jmm.0.001560. PMID 35771615
- [Derived] Bienvenu AL, Cour M, Pavese P, Guichon C, Leray V, Chapuis C, Dureault A, Mohkam K, Gallet S, Bourget S, Kahale E, Chaabane W, Subtil F, Maucort-Boulch D, Talbot F, Dode X, Richard JC, Leboucher G. Correlation between antifungal clinical practices and a new clinical decision support system ANTIFON-CLIC(R) for the treatment of invasive candidiasis: a retrospective multicentre study. J Antimicrob Chemother. 2024 Jun 3;79(6):1407-1412. doi: 10.1093/jac/dkae118. PMID 38656566